CLINICAL TRIAL: NCT07182513
Title: Turkish Version of the Hammersmith Neonatal Neurological Examination (HNNE) With High-Risk of Infants: A Study of Validity and Reliability
Brief Title: Turkish Version of the Hammersmith Neonatal Neurological Examination (HNNE)
Acronym: HNNE
Status: Recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: HNNE; UNIVERSİTY (Other: KAHRAMANMARAŞ SÜTÇÜ İMAM UNİVERSİTY)
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP); Infant ALL; Neurological Development; Neonatal
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: High-risk infants being followed in the NICU of the University Hospital's Faculty of Medicine will be included. A total of 120±10 high-risk infants will be included in the study, representing 10 times the number of items in the HNNE short version. Infants with high risk of CP: Periventricular hemorrhage, intracranial hemorrhage grade 2, 3, 4, cystic PVL, stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterus), perinatal stroke, perinatal asphyxia, RDS, BPD and infants receiving long-term O₂ support, sepsis due to gram-negative bacteria, NEC, infantile apnea, those with a low 5th minute Apgar score (3 and below), those diagnosed with intrauterine growth retardation, multiple births (twins, triplets), preterm infants with ROP, infants with prolonged severe hypoglycemia and hypocalcemia, infants who are SGA or LGA, infants receiving mechanical ventilation for more than 24 hours, infants born less than 32 weeks of gestation and weighing less than 1500 g.

SUMMARY:
High-risk infants are defined as an infant with a history of adverse environmental and biological factors that may lead to neuromotor developmental problems. This group includes premature babies born at less than 37 weeks, term babies with low birth weight (LBW), or babies with developmental delays due to various reasons. These babies are also monitored for cerebral palsy (CP). CP is the most common physical disability in childhood, with an incidence of 2.1 per 1000 births. CP encompasses a group of permanent impairments in movement and posture development resulting from injury to the developing brain. Thanks to preventive measures and advances in obstetric and neonatal care, the incidence and severity of CP are currently decreasing in some countries, and it is emphasized that recovery can be more rapid with the use of early diagnosis guidelines or protocols in follow-up units. Early detection and monitoring of infants in the community for CP is essential only with appropriate, valid, and reliable tools to minimize potential sequelae through the timely implementation of CP-specific interventions. International guidelines require monitoring of infants at high risk of CP. This follow-up should be conducted by an interdisciplinary team, including a neonatologist, pediatrician, pediatric neurologist, pediatric physiotherapist, speech-language-swallowing therapist, and special education specialist. Pediatric physiotherapists are an important part of this team for developmental follow-up and rehabilitation. The Hammersmith Neonatal Neurological Examination (HNNE) is a method developed by Dubowitz and used in both clinical and research neurological examinations of preterm and term infants, is the neonatal form of the Hammersmith Infant Neurological Examination (HINE). Its use in the Neonatal Intensive Care Unit (NICU) is crucial for beginning risk assessment as early as possible. Research has determined the optimality score for this test for term infants evaluated in the first days after birth. Subsequently, the current version of the HNNE was standardized by evaluating low-risk term and high-risk preterm infants (25-34 weeks) at term ages, 6-48 hours after birth.The aim of this study was to develop a Turkish version of the HNNE for high-risk infants in Turkey and determine its validity and reliability. The translated HNNE version, which was found to be valid and reliable in this population, will be suitable for use by all healthcare professionals in Turkey. This study also aimed to determine the predictive value of HNNE at corrected 3-4/6 and 12 months when used in the follow-up of at-risk infants in NICUs in Turkey.The study consists of two phases. The first phase consisted of translating the short version of the survey into Turkish and conducting its cultural adaptation. The second phase involved reliability analysis. The principles of Guillemin et al. and Beaton et al. will be used in the translation and cultural adaptation processes.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with periventricular hemorrhage, intracranial hemorrhage grades 2, 3, or 4, cystic periventricular leukomalacia (PVL), stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterus), perinatal stroke, perinatal asphyxia, and hydrocephalus.
2. Infants with chronic lung disease, respiratory lung disease (RDS), bronchopulmonary dysplasia (BPD), and long-term oxygen supplementation.
3. Preterm infants with sepsis due to gram-negative bacteria, necrotizing enterocolitis (NEC), and infantile apnea.
4. Preterm infants with a low 5-minute Apgar score (3 or below), diagnosed with intrauterine growth restriction, multiple births (twins, triplets), and preterm infants with Retinopathy of Prematurity (ROP).
5. Infants with prolonged severe hypoglycemia and hypocalcemia.
6. Babies who are small for gestational age (SGA), less than the 3rd percentile, or large for gestational age (LGA), greater than the 97th percentile.
7. Babies receiving mechanical ventilation for more than 24 hours.
8. Babies born at less than 32 weeks' gestation and weighing less than 1500 grams.

Exclusion Criteria:

1. Babies with congenital malformations (spina bifida, congenital muscular torticollis, arthrogryposis multiplex congenita, etc.)
2. Babies diagnosed with metabolic and genetic diseases (Down syndrome, spinal muscular atrophy, Duchenne muscular dystrophy, etc.)
3. Babies still intubated and mechanically ventilated at 3 months postterm

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal infants at term equivalent age (TEA) of 37-42 weeks with high risk of cerebral palsy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Hammersmith Neonatal Neurological Examination (HNNE) | one assessment at the term equivalent age (37-40 weeks)
  The HNNE consists of a standard 34-item proforma. Each item is numbered 3 to 5. These items are scored from 1 to 3. When an item falls between two columns, it is assigned the appropriate half-score within the columns (e.g., items scored between 2 and 3 receive 2.5 points; items scored between 1 and 2 receive 1.5 points). High scores indicate good neurological status.The items in this proforma are; It is divided into six categories: tone (10), tone patterns (5), reflexes (6), movements (3), abnormal symptoms (3), and behavior (7). The scores from these subsections are summed to create an optimality score for preterm and term infants. The short version of the scale consists of 12 items (12,13). The short HNNM scale will be scored by a physical therapist on all high-risk infants in the NICU, using a fixed tripod and video recording in an environment away from stimuli.HNNE wıll be scored 4 times for test-retest and inter-observer reliability.

SECONDARY OUTCOMES:
Demographic form | one assessment at term equivalent age (37-40 weeks)
  It will consist of a form that includes prenatal and postnatal risk factors of all infants, demographic information of infants and parents, and neurological evaluation, cranial US and MRI results of infants, if any.
Pretchl's General Movements (GMs) Assessment | 2 assessments (first at writing term age (from birth to 47 weeks), second at fidgety term age (49-60 weeks)
  Heinz Prechtl demonstrated the validity and reliability of this method by determining that infants without fidgety movements (FMs) at 3-5 months of age are at increased risk of developing CP. GMs assessment is performed at three stages: preterm, writhing, and fidgety.According to the Prechtl method, abnormal movements during the preterm and writhing stages are classified as poor repertoire (PR), cramped synchronized (CS), and chaotic (Ch) GMs.During this period, fidgety movements are scored as F+, absent (F-) or abnormal (AF).
Hammersmith Infant Neurological Examination | 3, 6, 9 and 12 months of age (4 times)
  It is administered to analyze the risk of neurological anomalies in preterm and term infants. This test is known to be a prognostic battery for identifying neural disorders in infants between 2 and 24 months postnatally. The HINM consists of a total of 37 items, divided into three sections: neurological examination, developmental motor milestones, and behavioral status. Administration time is 5-10 minutes. Optimization scores for infants aged 3 to 18 months are based on the frequency distribution of neurological findings in the population in that age group. An item is considered optimal when present in at least 90% of infants. Use of the HINM test's optimality score and cut-off scores for CP at 3, 6, 9, 12, and 24 months provides prognostic information regarding the level of motor development.The HINE will be applied to all babies at 3, 6, 9 and 12 months and the cut-off scores for CP will be interpreted.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Proffessor, Study Chair — Gazi University; Hatice adıgüzel tat, Associate Proffessor, Principal Investigator — Kahramanmaras Sutcu Imam University; Sadık Yurttutan, Proffessor, Study Chair — Kahramanmaras Sutcu Imam University; Hidayet Cuhaoğlu, Lecturer, Study Chair — Kastamonu University; Halil İbrahim Celik, Associate Proffessor, Study Chair — Bilge Çocuk Special Education and Rehabilitation Center
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No